CLINICAL TRIAL: NCT01727089
Title: A Phase II Study of Bevacizumab Alone or in Combination With TRC105 for Advanced Renal Cell Cancer
Brief Title: Bevacizumab With or Without TRC105 in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02206; NCI-2012-02206 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-121; PhII-121 (Other: City of Hope Comprehensive Cancer Center); 9144 (Other: CTEP); N01CM00038 (NIH); N01CM00039 (NIH); N01CM00071 (NIH); N01CM00099 (NIH); P30CA033572 (NIH)
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Carcinoma; Stage IV Renal Cell Cancer; Type 1 Papillary Renal Cell Carcinoma; Type 2 Papillary Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — carotuximab; Bevacizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (bevacizumab) (Active Comparator): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis
- Arm II (bevacizumab, anti-endoglin monoclonal antibody TRC105) (Experimental): Patients receive bevacizumab as in Arm I and anti-endoglin monoclonal antibody TRC105 IV over 1-4 hours on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-Endoglin Chimeric Monoclonal Antibody TRC105; Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Biological: Anti-Endoglin Chimeric Monoclonal Antibody TRC105 — Given IV
  Other Names: TRC105
  Arms: Arm II (bevacizumab, anti-endoglin monoclonal antibody TRC105)
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
  Arms: Arm II (bevacizumab, anti-endoglin monoclonal antibody TRC105)

SUMMARY:
This randomized phase II trial studies how well bevacizumab with or without anti-endoglin monoclonal antibody TRC105 (TRC105) works in treating patients with kidney cancer that has spread to other parts of the body (metastatic). Monoclonal antibodies, such as bevacizumab and anti-endoglin monoclonal antibody TRC105, may block tumor growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression-free survival at 12 and 24 weeks for bevacizumab alone or in combination with TRC105 (anti-endoglin monoclonal antibody TRC105).

SECONDARY OBJECTIVES:

I. Toxicity and Response Evaluation Criteria in Solid Tumors (RECIST) response rate for the combination compared to single agent bevacizumab.

TERTIARY OBJECTIVES:

I. To evaluate tumor tissue expression of endoglin (CD105), transforming growth factor, beta receptor II (TGFBR2), activin A receptor type II-like 1 (ACVRL1) and transforming growth factor, beta receptor 1 (TGFBR1) kinase from pre- and post-treatment tissue samples in order to determine whether CD105 and stem cell activation occurs after exposure to anti-vascular endothelial growth factor (VEGF) therapy as predicted by laboratory models, and whether exposure to anti-endoglin monoclonal antibody TRC105 affects these changes.

II. To compare the soluble CD105 levels at baseline and after treatment between the group receiving bevacizumab alone and the group receiving bevacizumab in combination with anti-endoglin monoclonal antibody TRC105.

III. To compare TGFBR2 levels at baseline and after treatment between the group receiving bevacizumab alone and the group receiving bevacizumab in combination with anti-endoglin monoclonal antibody TRC105.

IV. To evaluate whether circulating tumor cells (CTCs) can be detected in this patient population using parylene membrane filter technology, and whether changes in CTC counts and CD105 expression on CTCs during therapy correspond to imaging and clinical response.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15.

ARM II: Patients receive bevacizumab as in Arm I and anti-endoglin monoclonal antibody TRC105 IV over 1-4 hours on days 1, 8, 15, and 22.

In both arms, treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed renal cancer; all histologic subtypes will be eligible
* Patients must have metastatic disease which is measurable, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) to >= 20 mm in the long axis by chest x-ray, >= 10 mm in the long axis by spiral computed tomography (CT), magnetic resonance imaging (MRI), calipers, or clinical exam, or >= 15 mm in the short axis for lymph nodes
* Patients must have received at least 1 prior systemic therapy for renal cancer but no more than 4 prior therapies; they must have documented intolerance to or progression despite at least 1 systemic therapy; therapy administered in the adjuvant setting counts toward the prior systemic therapy total; if adjuvant therapy is the patient's only prior therapy the disease must have recurred during treatment or within 3 months of discontinuation
* Allowable prior therapies include VEGF tyrosine kinase inhibitor (TKIs), mammalian target of rapamycin (mTOR) inhibitors, and cytokine therapy (example: interleukin-2 [IL2])
* At least 2 weeks must have elapsed from the last dose of the prior systemic therapy for biologics and 4 weeks for chemotherapy (6 weeks for nitrosoureas or mitomycin C); also note that at least 3 weeks should have elapsed since prior TKI administration
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy of greater than 6 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< institutional upper limits or normal (except for Gilbert's)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal (except subjects with liver metastases, who can have AST/ALT =< 5 x ULN)
* Creatinine glomerular filtration rate (GFR) (calculated or measured) > 50 mL/min
* Hemoglobin >= 9 g/dL
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of TRC105 or bevacizumab administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had systemic biologic therapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events related to their prior therapy
* Patients who have previously been treated with bevacizumab
* Patients who have previously been treated with TRC105
* Patients who are receiving any other investigational agents
* Known central nervous system (CNS) disease except for treated brain metastasis; treated brain metastases are defined as having no ongoing requirement for steroids and no evidence of progression or hemorrhage after treatment for at least 3 months, as ascertained by clinical examination and brain imaging (MRI or CT) (stable dose of anticonvulsants are allowed); treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; gamma knife, linear accelerator [LINAC], or equivalent) or a combination as deemed appropriate by the treating physician; patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to day 1 will be excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TRC105 or bevacizumab
* Patients on full-dose anticoagulation will be excluded; antiplatelet therapy will not be exclusionary
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unhealed wound, gastrointestinal fistula, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction, cerebrovascular accident
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother wishes to participate in the study
* Patients with a history of bleeding diathesis or inherited coagulopathy are excluded; in addition, those with a history of deep vein thrombosis (DVT) or pulmonary embolus within 1 year and still requiring active anticoagulation will be excluded; those with a more remote history of DVT or pulmonary embolus may be eligible but the risk of recurrent thrombosis should be considered
* Patients with history of hereditary hemorrhagic telangiectasis (HHT-1 and HHT-2)
* Serious or non-healing wound, ulcer, or bone fracture OR history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to day 1
* Invasive procedures defined as follows:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to day 1 therapy
  * Anticipation of need for major surgical procedures during the course of the study
  * Core biopsy within 7 days prior to day 1 therapy
* Patients with clinically significant cardiovascular disease are excluded:

  * Inadequately controlled hypertension (HTN) (systolic blood pressure [SBP] > 160 mmHg and/or diastolic blood pressure [DBP] > 90 mmHg despite antihypertensive medication)
  * History of cerebrovascular accident (CVA) within 6 months
  * Myocardial infarction or unstable angina within 6 months
  * New York Heart Association grade II or greater congestive heart failure
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g. aortic aneurysm, history of aortic dissection)
  * Clinically significant peripheral vascular disease
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Patients with psychiatric illness/social situations that would limit compliance with study requirements will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Dorff, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (30):
- United States (28):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado, Denver, Colorado
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc - Jefferson Boulevard, Fort Wayne, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia
- National Taiwan University Hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Bevacizumab): Patients receive 10 mg/kg bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Bevacizumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
- Arm II (Bevacizumab, Anti-endoglin Monoclonal Antibody TRC105): Patients receive 10 mg\kg bevacizumab as in Arm I and anti-endoglin monoclonal antibody TRC105 10 mg\kg IV over 1-4 hours on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Anti-Endoglin Chimeric Monoclonal Antibody TRC105: Given IV
  Bevacizumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
Period: Overall Study
Arm/Group | Arm I (Bevacizumab) | Arm II (Bevacizumab, Anti-endoglin Monoclonal Antibody TRC105)
Started | 29 | 30
Completed | 29 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Bevacizumab) | Arm II (Bevacizumab, Anti-endoglin Monoclonal Antibody TRC105) | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Median (Full Range); unit: years] | 58 [25 to 82] | 65 [24 to 78] | 60 [24 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 20 | 24 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 22 | 27 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 24 | 28 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 24 Weeks
Description: Progression-free survival 24 after starting treatment. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: The duration of time from start of treatment to time of progression or death, assessed at 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Bevacizumab) | Arm II (Bevacizumab, Anti-endoglin Monoclonal Antibody TRC105)
Number analyzed (Participants) | 29 | 30
percentage of participants | 52 [36 to 76] | 27 [15 to 50]

2. Primary Outcome: Progression-free Survival at 12 Weeks
Description: Progression-free survival 12 after starting treatment. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: The duration of time from start of treatment to time of progression or death, assessed at 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Bevacizumab) | Arm II (Bevacizumab, Anti-endoglin Monoclonal Antibody TRC105)
Number analyzed (Participants) | 29 | 30
percentage of participants | 66 [51 to 86] | 58 [42 to 71]

3. Secondary Outcome: Number of Participants With Grade 3 and Above Adverse Events (AE) Related to Treatment
Description: The descriptions and grading scales found in the revised National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 will be utilized for AE reporting.
  Grade 1 - Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 - Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL).
  Grade 3 - Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  Grade 4 - Life-threatening consequences; urgent intervention indicated. Grade 5 - Death related adverse event.
Time Frame: From time of treatment initiation until 30 days post treatment, assessed every 4 weeks.
Measure: Number; unit: participants
Arm/Group | Arm I (Bevacizumab) | Arm II (Bevacizumab, Anti-endoglin Monoclonal Antibody TRC105)
Number analyzed (Participants) | 29 | 30
participants
  Abdominal pain | 3 | 3
  Anemia | 4 | 8
  Anorexia | 0 | 1
  Bleeding | 2 | 0
  bronchopulmonary hemorrhage | 1 | 0
  Fatigue | 0 | 2
  Hypercalcemia | 0 | 2
  Hypertension | 5 | 4
  Hyponatremia | 1 | 2
  Infusion reaction | 0 | 2
  Nausea/vomitting | 0 | 5
  Proteinuria | 2 | 0

4. Secondary Outcome: Number of Participants With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: From time of treatment initiation until conclusion of treatment, assessed every 12 weeks.
Measure: Number; unit: participants
Arm/Group | Arm I (Bevacizumab) | Arm II (Bevacizumab, Anti-endoglin Monoclonal Antibody TRC105)
Number analyzed (Participants) | 29 | 30
participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 2 years and 7 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Arm I (Bevacizumab) | Arm II (Bevacizumab, Anti-endoglin Monoclonal Antibody TRC105)
All-Cause Mortality (participants affected / at risk) | 4/29 | 5/30
Serious Adverse Events (participants affected / at risk) | 10/29 | 14/30
Other Adverse Events (participants affected / at risk) | 29/29 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Bevacizumab) (N=29) | Arm II (Bevacizumab, Anti-endoglin Monoclonal Antibody TRC105) (N=30)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 2 (3) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (2) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Death NOS (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Failure to thrive (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Fever (General disorders) | 1 (2) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Weakness (General disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2)
progression of renal cell cancer (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Grade 5, possibly related
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
scalp laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (13)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Bevacizumab) (N=29) | Arm II (Bevacizumab, Anti-endoglin Monoclonal Antibody TRC105) (N=30)
Anemia (Blood and lymphatic system disorders) | 10 (29) | 16 (79)
Sinus bradycardia (Cardiac disorders) | 3 (11) | 5 (9)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 5 (13)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 2 (2)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Itchy Eyes (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
suconjunctival hemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (3) | 2 (6)
Abdominal pain (Gastrointestinal disorders) | 8 (11) | 4 (14)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (3) | 1 (1)
Blood in Stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (13) | 8 (10)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 2 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (9) | 10 (16)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (17)
Oral pain (Gastrointestinal disorders) | 1 (2) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal discharge (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue Ulcerations (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 7 (9)
diverticulosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
hiatal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloody Gums (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 4 (6) | 2 (5)
Cracked Lips (General disorders) | 0 (0) | 1 (1)
Death NOS (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 4 (4) | 5 (6)
Fatigue (General disorders) | 18 (54) | 23 (79)
Fever (General disorders) | 4 (5) | 3 (3)
Flu like symptoms (General disorders) | 1 (1) | 1 (1)
Increased Thirst (General disorders) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 5 (6)
Localized edema (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Night sweats (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (4)
Pain (General disorders) | 2 (7) | 7 (11)
Rash (General disorders) | 0 (0) | 1 (1)
Swelling of Feet (General disorders) | 0 (0) | 1 (1)
swelling of feet (General disorders) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 3 (4)
Upper respiratory infection (Infections and infestations) | 1 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (14)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Activated partial thromboplastin time pr (Investigations) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (26) | 3 (5)
Alkaline phosphatase increased (Investigations) | 7 (13) | 6 (11)
Aspartate aminotransferase increased (Investigations) | 6 (17) | 7 (9)
Blood bilirubin increased (Investigations) | 1 (1) | 3 (3)
Cardiac troponin T increased (Investigations) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 1 (2) | 0 (0)
Creatinine increased (Investigations) | 7 (15) | 6 (14)
Elevated BUN (Investigations) | 2 (2) | 0 (0)
Elevated BUN count (Investigations) | 1 (1) | 0 (0)
Elevated Eos Auto (Investigations) | 1 (1) | 0 (0)
Elevated LDH (Investigations) | 1 (3) | 0 (0)
GGT increased (Investigations) | 1 (6) | 0 (0)
Hemoglobin increased (Investigations) | 1 (6) | 0 (0)
INCREASED LDH (Investigations) | 1 (3) | 0 (0)
INR increased (Investigations) | 1 (3) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Low Co2 (Investigations) | 0 (0) | 1 (2)
Low LDH (Investigations) | 1 (2) | 0 (0)
Low chloride count (Investigations) | 1 (3) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 4 (7)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 6 (22) | 3 (4)
Weight gain (Investigations) | 2 (3) | 5 (22)
Weight loss (Investigations) | 3 (7) | 4 (9)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
creatinine increased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 9 (19) | 9 (15)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 7 (8)
GLUCOSURIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (7) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (18) | 8 (35)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (16) | 9 (13)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 3 (6) | 4 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (21) | 8 (28)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (5) | 4 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (7) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 11 (25) | 11 (29)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 3 (5) | 3 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 7 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (7)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Intermittent Chest Wall Tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (7) | 3 (3)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
anterolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
lumbar disk degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (7) | 5 (10)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 10 (22) | 15 (25)
Lethargy (Nervous system disorders) | 0 (0) | 1 (2)
Paresthesia (Nervous system disorders) | 1 (2) | 2 (4)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (3) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Rigors (Nervous system disorders) | 0 (0) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1) | 1 (9)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2) | 3 (3)
Confusion (Psychiatric disorders) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4)
Burning sensation in urine (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 4 (8) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyaline casts >2 (Renal and urinary disorders) | 1 (1) | 0 (0)
Leukocyte Esterase 3+ (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 11 (43) | 8 (20)
RBC's > 50 (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary fistula (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (3) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
WBC's > 50 (Renal and urinary disorders) | 1 (1) | 0 (0)
pneumaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Bradypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 7 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 9 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 16 (56)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 3 (7)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (7)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
nose bleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ABRASION LEFT HAND (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Face and Scalp Skin Lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Face and scalp lesions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Neck rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndro (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (33)
Rash on face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Tenderness/Redness on Hands (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
cold sores (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
inflamed skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
pallor (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
redness of palm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
skin reddened (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
skin redness: palm (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hair thinning (Social circumstances) | 1 (1) | 0 (0)
Port-A-Cath insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 6 (10)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 17 (50) | 15 (55)
Hypotension (Vascular disorders) | 3 (3) | 6 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT01727089/Prot_SAP_000.pdf